CLINICAL TRIAL: NCT00755001
Title: Clinical Study on BiHapro Total Hip System With Different Surface Coatings
Status: Terminated | Type: Observational
Why Stopped: The site decided to stop the study
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet Spain Orthopaedics S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: BMET EP 01
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Osteoarthritis
Keywords: Total Hip Replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with Plasma HA: BiHapro Hip stem with PPS Ti + Plasma HA
  Interventions: Device: BiHapro hip stem with PPS Ti+Plasma HA
- with BoneMaster HA: BiHapro Hip stem with PPS Ti + BoneMaster HA
  Interventions: Device: BiHapro hip stem with PPS Ti+BoneMaster HA

INTERVENTIONS:
Device: BiHapro hip stem with PPS Ti+Plasma HA — BiHapro hip stem with PPS Ti+Plasma HA
  Other Names: BiHapro hip stem
  Groups: with Plasma HA
Device: BiHapro hip stem with PPS Ti+BoneMaster HA — BiHapro hip stem with PPS Ti+BoneMaster HA
  Other Names: BiHapro hip stem
  Groups: with BoneMaster HA

SUMMARY:
This post market study intends to evaluate the safety and the performance of BiHapro Total Hip System with two types of coatings.

DETAILED DESCRIPTION:
The efficacy of the prosthesis will be evaluated comparing the pain, the function and the range of motion measured preoperatively and postoperatively using recognized clinical outcomes Harris Hip Score. The secondary efficacy measurement is based on X-rays to measure the mineral bony thickness in the areas of Gruen zones of the proximal femur.

ELIGIBILITY:
The patients who are selected for this study must fit the following criteria.

* Candidate for a Total Hip Arthroplasty
* Less than 80 years of age.
* A pre-operative level of pain and function the same as for conventional joint replacement.
* A likelihood of obtaining relief of pain and improved function.
* Full skeletal maturity.
* Ability to follow instructions.
* Good general health for age.
* Willing to return for follow-up evaluations.
* No bias to sex.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Total Hip Arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | annual at least to 5 yr

SECONDARY OUTCOMES:
Radiographic Assessment | Annual; At least to 5 yr

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - University Hospital of Aviles, Avilés
  - University Central Hospital of Asturias, Oviedo